CLINICAL TRIAL: NCT01223989
Title: Evaluation of the Utility of an Hypocaloric Diet With or Without Bread in Overweight/Obesity Treatment
Brief Title: Bread in Overweight/Obesity Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Carmen Gómez Candela, Fundacion para la Investigacion Biomedica del Hospital La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP 753
Record Dates: First submitted 2010-10-13; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; bread; hypocaloric diet
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group bread (Experimental): group who received an hypocaloric balanced diet including bread
  Interventions: Other: hypocaloric diet balanced + nutrition education + ruled physical activity
- group without bread (Active Comparator): group who received a hypocaloric balanced diet with exclusion of bread
  Interventions: Other: hypocaloric diet balanced + nutrition education + ruled physical activity

INTERVENTIONS:
Other: hypocaloric diet balanced + nutrition education + ruled physical activity

SUMMARY:
The purpose of this study is to determine the utility of an hypocaloric diet with or without bread in patients with overweight and obesity

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* sex female
* signed informed consent
* patient with overweight and obesity (IMC: > 25 < 39.9)

Exclusion Criteria:

* Family and social environment that prevents compliance with treatment diet.
* Having to perform any kind of diet special sickness associated: Celiac disease, chronic renal failure, etc.
* patients with Diabetes Mellitus.
* patients with Eating disorders.
* patients with Dementia, Mental illness or impaired function cognitive.
* consuming drugs or substances for losing weight (except in those cases in which suspension thereof 15 days of beginning the study).
* Present disease which may interfere with weight loss: serious psychiatric disease, hypothyroidism not controlled.
* Be pregnant or period of lactation.
* Inability to comply with the physical activity plan agreed.
* Want to quit smoking during the time that lasts for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
changes in anthropometric parameters | after 16 weeks of start the diet
  weight, height, BMI, fat mass, lean mass.

SECONDARY OUTCOMES:
changes in biochemical parameters | after 16 weeks of start the diet
  hematocrit, hemoglobin, lipid profile, ghrelin, leptin, adiponectin.
Adherence | after 16 weeks of start the diet
  Validated scale
change in satiety and hunger Test | after 16 weeks of start the diet
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Gómez Candela, PhD, Principal Investigator — Jefe Unidad Nutrición Clínica y Dietética Hospital Universitario La Paz

REFERENCES:
- [Derived] Loria-Kohen V, Gomez-Candela C, Fernandez-Fernandez C, Perez-Torres A, Garcia-Puig J, Bermejo LM. Evaluation of the usefulness of a low-calorie diet with or without bread in the treatment of overweight/obesity. Clin Nutr. 2012 Aug;31(4):455-61. doi: 10.1016/j.clnu.2011.12.002. Epub 2011 Dec 30. PMID 22209501